CLINICAL TRIAL: NCT00882635
Title: The STrategic Reperfusion Early After Myocardial Infarction (STREAM) Anticoagulation With Enoxaparin vs. Unfractionated Heparin in Primary PCI Sub-study.
Brief Title: The STREAM Percutaneous Coronary Intervention Anticoagulant Sub-study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Robert Welsh (Other)
Collaborators: Sanofi (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Robert Welsh, Associate Professor, University of Alberta
Organization: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STREAMPCI
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI; acute coronary syndromes; primary percutaneous coronary intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Acute Coronary Syndrome | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enoxaparin (Experimental)
  Interventions: Drug: enoxaparin
- Unfractionated heparin (Active Comparator)
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: enoxaparin — Enoxaparin 0.5 mg/kg IV bolus (Regardless of whether the investigator has chosen to initiate concomitant GP IIb/IIIa antagonist; provision for additional IV enoxaparin to be administered if elapsed time to PCI exceeds 2 hours (from original IV dose) - enoxaparin 0.25 mg/kg IV will be administered At the discretion of the treating physician, if sustained anticoagulation is required then enoxaparin subcutaneously will be administered - enoxaparin 1.0 mg/kg SQ q 12 hours.
  Maintenance dose adjustment for renal insufficiency - creatinine clearance < 30 ml/min, sc enoxaparin should be administered at 1.0 mg / kg / q24 hours. No adjustment of IV dose is required in case of renal insufficiency
  Arms: Enoxaparin
Drug: Unfractionated heparin — Unfractionated heparin 70 u/kg IV bolus (consistent with ASSENT 4 PCI) Baseline ACT will be draw at time of sheath insertion - With use of GP IIb/IIIa antagonist additional UFH will be administered to achieve an ACT of ≥200 - 250 seconds If IIb/IIIa is not utilized - additional UFH will be administered to achieve an ACT of ≥250-350 seconds At the discretion of the treating physician if sustained anticoagulation is required:UFH infusion 12/u/kg/hr IV infusion to commence
  Arms: Unfractionated heparin

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Enoxaparin and Unfractionated Heparin in St Elevation Myocardial Infarction patients undergoing primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
Past research in stable patients with coronary artery disease and those with non-ST elevation acute coronary syndromes (NSTEMI) has demonstrated the safety and efficacy of enoxaparin as an anticoagulant strategy in patients undergoing percutaneous coronary intervention 1-3.

In patients with ST-elevations myocardial infarction (STEMI) receiving pharmacological reperfusion (fibrinolysis), enoxaparin has been shown to be an attractive alternative to unfractionated heparin based upon past modest scale trials (HART-2, ENTIRE TIMI 23, ASSENT-3, ASSENT-3+)4-6. These results were definitively extended by the ExTRACT-TIMI 25 trial which compared fibrinolysis with unfractionated heparin versus enoxaparin in 20,506 patients with STEMI 7. The primary endpoint of death and re-MI occurred in 9.9% of patients with enoxaparin and 12.0% of patients in the unfractionated heparin group (17% RR, p<0.001); major bleeding occurred in 2.1% and 1.4% respectively (p<0.001). This was achieved using a dose reduction strategy in the elderly (>75yrs) that omitted the intravenous enoxaparin bolus and decreased the subcutaneous injection to 0.75 mg/kg. After initial fibrinolysis, fewer patients underwent PCI through 30 days in the enoxaparin group versus the unfractionated heparin group (22.8% vs 24.2%, p=0.027). Among those who underwent PCI (n=4674) by 30 days the primary endpoint occurred in 10.7% with enoxaparin versus 13.8% unfractionated heparin randomization (0.77 RR, p<0.001); major bleeding was not different (1.4% vs. 1.6%, p=NS) 8.

Despite existing data in stable coronary artery disease, NSTEMI, and STEMI patients treated with fibrinolysis there is limited data regarding the approach to anticoagulation therapy with enoxaparin in those STEMI patients undergoing primary PCI. Within a sub-study of the Which Early ST Elevation Myocardial Infarction Therapy study (WEST) we undertook systematic anti-Xa sampling to address the adequacy of anticoagulation with an enoxaparin based regime9, 10. WEST patients undergoing primary PCI received aspirin, clopidogrel, and subcutaneous enoxaparin (1mg/kg) at the time of randomization. Subsequent administration of intravenous enoxaparin and abciximab at the time of PCI was encouraged. Those receiving supplemental intravenous enoxaparin (0.3 - 0.5 mg/kg) in addition to subcutaneous enoxaparin achieved anti-Xa levels > 0.5 units/ml (the proposed therapeutic concentration). Amongst those receiving 1 mg/kg of enoxaparin subcutaneous at randomization and 0.3 mg/kg intravenous enoxaparin at time of PCI, none had excessive anticoagulation (anti-Xa > 1.5 units/ml) suggesting that this may be an attractive dosing strategy.

Recently a non-randomized comparison of unfractionated heparin and enoxaparin within the FINNESSE study was presented in STEMI patients undergoing primary PCI. Preliminary reports indicate superior outcomes amongst those receiving enoxaparin 0.5mg/kg intravenous as compared to unfractionated heparin intravenously.

The STREAM study provides a unique and important opportunity to acquire randomized safety and efficacy data on anticoagulation with enoxaparin vs. unfractionated heparin in STEMI patients undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal or greater than 18 years
2. Onset of symptoms of STEMI < 3 hours prior to randomisation
3. 12-lead ECG (ST elevation will be measured from the J point) indicative of an acute STEMI: >2 mm ST elevation across 2 contiguous precordial leads (best 2 of V1-V6) or leads I, AVL for a minimum combined total of >4 mm ST elevation,or >3 mm ST elevation in 2 contiguous inferior leads (best 2 of II, III, AVF) for a minimum combined total of > 6 mm ST elevation.
4. Informed consent received

Exclusion Criteria:

1. PCI (1st balloon inflation) expected to commence < 60 minutes from diagnosis (qualifying ECG) or inability to arrive at the cardiac catheterization laboratory (1st balloon inflation) within 3 hours after randomisation.
2. Anticipated or obvious problem with vascular access.
3. Previous CABG
4. Left bundle branch block or ventricular pacing.
5. Patients with cardiogenic shock - Killip Class 4
6. Patients with a body weight < 55 kg (known or estimated)
7. Uncontrolled hypertension, defined as blood pressure measurement > 180/110 mm Hg (systolic BP > 180 mm Hg and/or diastolic BP > 110 mm Hg) confirmed on repeat measures (2 documented measurements at any time) prior to randomization.
8. Known use oral anticoagulants (warfarin or coumadin) or GP IIb/IIIa antagonists within the preceding 7 days or recent administration of any IV or SC anticoagulation within 12 hours including: unfractionated heparin, enoxaparin, and/or bivalirudin.
9. Active bleeding, known bleeding diathesis/disorder including thrombocytopenia or clinical diagnosis associated with increased risk of bleeding including: known active peptic ulceration and/or neoplasm with increased bleeding risk.
10. Major surgery, biopsy of a parenchymal organ, or significant trauma within the past 2 months (this includes any trauma associated with the current AMI)
11. Any history of central nervous system abnormality (i.e. neoplasm, aneurysm, intracranial or spinal surgery) or recent trauma to the head or cranium (i.e <3 months)
12. Any known history of haemorrhagic stroke or stroke of unknown origin
13. Ischaemic stroke or transient ischaemic attack (TIA) in the preceding 6 months
14. Prolonged or traumatic cardiopulmonary resuscitation (> 10 minutes) within the past 2 weeks
15. Known acute pericarditis and/or subacute bacterial endocarditis
16. Known acute pancreatitis or known severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis
17. Chronic dialysis or known renal insufficiency (prior S-creatinine >2.5 mg% (>220 µmol/l) for men and >2.0 mg% (>175 µmol/l)) for women
18. Pregnancy or lactation or parturition within the previous 30 days; women of childbearing potential must be using a medically accepted method of birth control
19. Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 7 days
20. Known hypersensitivity to tenecteplase, alteplase, ASA, clopidogrel, enoxaparin, or to any of the excipients or to the contrast media used in angiography Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk if the investigational therapy is initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adequacy of anticoagulation with enoxaparin (anti-Xa levels ≥ 0.5 U/ml to 1.5 U/ml) vs. unfractionated heparin (ACT - ≥200 - 250 seconds with concomitant GP IIb/IIIa antagonist and ACT - ≥250 - 350 seconds without concomitant GP IIb/IIIa antagonist). | During Primary PCI

SECONDARY OUTCOMES:
Composite of major bleeding (non-CABG), death, cardiogenic shock, and congestive heart failure | 30 days
ECG & angiographic measures before and after primary PCI | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Welsh, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Southlake, Newmarket, Ontario